CLINICAL TRIAL: NCT07334626
Title: Impact of Pilates Exercises on Bone Mineral Density in Breast Cancer Survivors Receiving Hormonal Therapy
Acronym: PilatesBCS2026
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mahmoud Hamada Mohamed, Associate Professor of Physical Therapy, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pilates on osteoporosis BCS26
Record Dates: First submitted 2025-12-28; First posted 2026-01-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Breast Cancer Survivors; Aromatase Inhibitors; Osteoporosis or Osteopenia; Pilates Exercise
Keywords: pilates exercises; breast cancer survivors; bone mineral denisty; aromatase inhibitors
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis; Bone Diseases, Metabolic | interventions — Exercise Movement Techniques; Calcium

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant) This is a parallel group randomized controlled trial with two arms receiving different interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental)
  Interventions: Other: Pilates Exercises; Drug: Calcium and Vitamin D Supplementation
- Control group (Active Comparator)
  Interventions: Drug: Calcium and Vitamin D Supplementation

INTERVENTIONS:
Other: Pilates Exercises — The Pilates program will consist of mat-based exercises with optional use of light equipment such as resistance bands and small weights. Each session will last 60 minutes and will be performed three times per week over a total duration of 12 weeks. The program will follow a structured progression with systematic increases in exercise difficulty, load, and repetitions based on individual tolerance. The intervention will focus on enhancing core control, spinal extension and posture, lower-limb weight-bearing activities, and balance. Sessions will be initially supervised by a trained physiotherapist with expertise in oncology rehabilitation.
  Arms: Study group
Drug: Calcium and Vitamin D Supplementation — Participants will receive daily oral calcium supplementation at a total dose of 1,200 mg/day, combined with vitamin D (total daily vitamin D dose: 200 IU), administered throughout the study period as part of standard osteoporosis management for breast cancer survivors receiving hormonal therapy.

SUMMARY:
Breast cancer survivors receiving endocrine (hormonal) therapy (aromatase inhibitors) are at high risk for cancer treatment-induced bone loss and osteoporosis due to estrogen depletion.

DETAILED DESCRIPTION:
Pilates is a safe, low-impact exercise approach that may help manage osteoporosis in breast cancer survivors by improving postural control, core strength, balance, and functional mobility. When appropriately modified, Pilates supports musculoskeletal health, reduces fall risk, and promotes safe movement patterns, making it a suitable intervention for osteoporosis-focused clinical trials in this population.

Guidelines recommend weight-bearing and resistance exercise to slow bone loss, but no RCT has specifically tested Pilates for bone health outcomes in this population.

Existing trials have shown Pilates improves strength and balance, which are relevant for fracture risk, but bone mineral density (BMD) has not yet been clearly evaluated The aim of this study is to evaluate the effect of a 12-weeks Pilates program on bone mineral density (BMD) at the lumbar spine and hip in breast cancer survivors on hormonal therapy.

A total of 60 patients (n=30 per group). Breast cancer survivors receiving endocrine (hormonal) therapy ( aromatase inhibitors) in the past 3 months. Participants will be recruited from Benha University hospital and local oncology clinics in benha. Participants will be screened for eligibility prior to being enrolled in the study participating in the study assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Female breast cancer survivors aged 40-60 years.
2. Histologically confirmed stage I-III breast cancer.
3. Currently receiving hormonal therapy (aromatase inhibitors) for at least 3 months.
4. At risk of osteoporosis or with low bone mineral density (BMD) defined by T-score ≤ -1.0 at lumbar spine or hip.
5. Medically cleared for exercise, specifically low-to-moderate intensity Pilates.
6. Able to attend supervised exercise sessions three times per week for 12 weeks.
7. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Metastatic (stage IV) or recurrent breast cancer.
2. History of osteoporotic fractures in the past 12 months.
3. Severe cardiovascular, respiratory, or musculoskeletal conditions that contraindicate exercise.
4. Uncontrolled hypertension, diabetes, or thyroid disorders.
5. Current use of corticosteroids.
6. Active bone metabolic disease other than osteoporosis (e.g., Paget's disease, osteomalacia).
7. Severe cognitive impairment or psychiatric illness preventing adherence to exercise or supplementation.
8. Known allergy or intolerance to calcium or vitamin D supplementation.
9. Participation in another clinical trial with structured exercise or bone-targeted intervention within the last 3 months.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density (BMD) measurement | Base line and after 12 weeks
  Change in bone mineral density (BMD) at the lumbar spine and total hip (g/cm²) from baseline to 12 weeks. BMD will be measured using dual-energy X-ray absorptiometry (DEXA), which is the standard technique for assessing BMD at the lumbar spine and proximal femur. The BMD and T-score of the femoral neck and lumbar vertebrae will be determined using a Hologic Discovery W series DEXA scanner.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire. | Base line and after 12 weeks
  Change in health-related quality of life (HRQoL) from baseline to 12 weeks, assessed using the Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire. The FACT-B is a validated, self-administered instrument that evaluates five domains: physical well-being, social/family well-being, emotional well-being, functional well-being, and breast cancer-specific concerns. Scores for each domain and the total FACT-B score will be calculated according to standardized scoring guidelines, with higher scores indicating better quality of life. Participants will complete the questionnaire at baseline (pre-intervention) and at 12 weeks (post-intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinic, faculty of Physical Therapy, Benha university, Banhā, Benha, Egypt

IPD SHARING:
Plan to Share IPD: Undecided